CLINICAL TRIAL: NCT01334528
Title: Consistency of ANAM Performance in Those With Deployment Acquired Mild TBI
Brief Title: Consistency of Automated Neuropsychological Assessment Metrics (ANAM) Performance in Those With Deployment Acquired Mild Traumatic Brain Injury (TBI)
Acronym: ANAM
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Brenner, Director, VISN19 MIRECC, VA Eastern Colorado Health Care System
Other Study IDs: 10-1483
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Mild Traumatic Brain Injury; Post-Concussive Symptoms
Keywords: Deployment Acquired Mild Traumatic Brain Injury; Persistent Post-Concussive Symptoms; Repeated measures
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OEF/OIF Veterans mTBI: Operation Iraqi Freedom (OIF)/Operation Enduring Freedom (OEF) Veterans with a history of mild traumatic brain injury (mTBI) with persistent self-reported symptoms.

SUMMARY:
The purpose of this project is to explore the degree to which performance consistency on neuropsychological measures varies in a sample of Operation Iraqi Freedom (OIF)/Operation Enduring Freedom (OEF) Veterans with a history of mild traumatic brain injury (mTBI) with persistent self-reported symptoms.

DETAILED DESCRIPTION:
Mild TBI outcome studies are traditionally limited to single administration or baseline/post-injury assessment models and they often fail to show enduring deficits among persons complaining of such problems. It may be the case that our standard approach to deficit measurement in mTBI has confounded our ability to elicit the actual impairment. The proposed study could generate an assessment paradigm shift (performance over time) and afford professionals the direction to better assess and ultimately serve persons with mTBI. Additionally, research on the impact of PTSD symptoms on throughput and cognitive performance has been mixed (Bremner et al., 1995; Brenner et al, 2010; Vasterling et al., 1998, 2002, 2006) and the proposed study will yield additional data in that area.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45 years old
* At least one OEF/OIF deployment
* Currently receiving physical and/or mental health care through the VA Eastern Colorado Health Care System
* For TBI group - veteran must have a history of at least one deployment- related mild TBI with persistent symptoms

Exclusion Criteria:

* Effortful performance on the Test of Memory Malingering (TOMM)
* History of other significant neurological disease (other than mild TBI for the appropriate group) as assessed by interview and chart review
* History or diagnosis of deployment-related moderate or severe TBI or mild TBI without persistent symptoms for the TBI groups, or any history of deployment-related TBI for the non-TBI group, as assessed by interview and chart review
* History or diagnosis of non-deployment-related TBI
* Diagnosis of Schizophrenia or Bipolar Mood DisorderI Disorder as assessed by interview and/or chart review.
* Problematic drinking behavior that consistently exceeds recommended drinking limits per day, e.g., Diagnosis of Alcohol Abuse Disorder or Alcohol Dependence Disorder per the MINI; or five or more alcoholic drinks per day, four out of seven days per week for the previous two weeks or during the assessment process
* Use of illicit substance(s) more than five times in the two weeks before enrollment or during the testing process.
* Inability to read the informed consent document or adequately respond to questions regarding the informed consent procedure

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Operation Iraqi Freedom (OIF)/Operation Enduring Freedom (OEF) Veterans with a history of mild traumatic brain injury (mTBI) with persistent self-reported symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Automated Neuropsychological Assessment Metrics (v4; ANAM4™) | Over the course of 4 days
  The ANAM4™ Traumatic Brain Injury (TBI) Battery is a selection of tests from the ANAM4™ library (C-SHOP, 2007) believed to be especially sensitive to mild TBI. This battery was designed to aid in the assessment of general cognitive function following a suspected brain injury or other cognitive insult. The ANAM4 TBI battery includes the following tests: Simple Reaction Time, Procedural Reaction Time, Matching to Sample, Code Substitution-Learning, Code Substitution-Delayed Memory and Mathematical Processing and takes approximately 20 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, Ph.D., Principal Investigator — Eastern Colorado Health Sciences Denver VA MIRECC
Locations (1):
- Eastern Colorado Health Sciences Denver VA MIRECC, Denver, Colorado, United States

REFERENCES:
- See also: MIRECC of the VA Rocky Mountain Network (VSN 19) — http://www.mirecc.va.gov/visn19/index.asp